CLINICAL TRIAL: NCT03797768
Title: Protocol for Community-based Management of Chronic Obstructive Pulmonary Disease in Nepal: a Community-based Cluster Randomized Controlled Trial
Brief Title: Community-based Management of Chronic Obstructive Pulmonary Disease in Nepal
Acronym: COBIN-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AUTBA18
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Behavioural-FCHV Visit
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Behavioural-FCHV Visit — Female Community Health Volunteer will visit selected households on average 3 times a year for providing health promotion messages on improving lung health status and avoiding risk factors to COPD.
  Arms: Intervention

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the fourth most important cause of death worldwide and is one of the commonest non-communicable diseases (NCDs) in Nepal. The presence of risk factors like indoor and outdoor air pollution, the high prevalence of smoking and lack of general awareness of COPD makes it a serious public health concern. However, no attempt has been made in Nepal to estimate its burden and address the disease at the community level. This community-based cluster randomized controlled study aims to fulfil that gap through mobilization of Female Community Health Workers (FCHVs) who will be trained to perform a certain set of health promotion activities aimed at prevention of the disease and its progression. Baseline and follow-up surveys will be conducted to compare the intervention and control groups. This study has the potential to generate evidence in helping address NCDs in Nepal and also other similar resource-limited countries.

ELIGIBILITY:
Inclusion Criteria:

* Capable of performing spirometry
* Aged greater than and equal to 40 years
* Full time residents in the study area and will be in the study area for at least one year

Exclusion Criteria:

* Younger than 40 years of age
* Self-reported pregnancy
* having active pulmonary tuberculosis or being on medications for pulmonary tuberculosis
* thoracic, abdominal or eye surgery in the last six months
* History of Mental illness
* MI in past 8 weeks prior to study
* Hospital admission in the past six months for cardiac illness
* Those who decline to provide consent to the study will be excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1438 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second | 1 year
  Mean difference in FVE1 between intervention and control arm

SECONDARY OUTCOMES:
Proportion of risk factors of COPD between intervention and control arm | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tara Ballav Adhikari, MScPH, Principal Investigator — Department of Public Health, Aarhus University, Aarhus, Denmark
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari TB, Acharya P, Hogman M, Neupane D, Karki A, Drews A, Cooper BG, Sigsgaard T, Kallestrup P. Prevalence of Chronic Obstructive Pulmonary Disease and its Associated Factors in Nepal: Findings from a Community-based Household Survey. Int J Chron Obstruct Pulmon Dis. 2020 Sep 29;15:2319-2331. doi: 10.2147/COPD.S268110. eCollection 2020. PMID 33061350
- [Derived] Adhikari TB, Neupane D, Karki A, Drews A, Cooper B, Hogman M, Sigsgaard T, Kallestrup P. Community-based intervention for prevention and management of chronic obstructive pulmonary disease in Nepal (COBIN-P trial): study protocol for a cluster-randomized controlled trial. Trials. 2021 Jul 21;22(1):474. doi: 10.1186/s13063-021-05447-7. PMID 34289879
- See also: Prevalence of Chronic Obstructive Pulmonary Disease and its Associated Factors in Nepal: Findings from a Community-based Household Survey — https://doi.org/10.2147/COPD.S268110